CLINICAL TRIAL: NCT04893109
Title: A Randomized Phase II Trial of Adjuvant Trastuzumab Emtansine (T-DM1) Followed by Subcutaneous Trastuzumab Versus Paclitaxel in Combination With Subcutaneous Trastuzumab for Stage I HER2-positive Breast Cancer (ATEMPT 2.0)
Brief Title: ATEMPT 2.0: Adjuvant T-DM1 vs TH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Sara Tolaney, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-159
Record Dates: First submitted 2021-05-07; First posted 2021-05-19 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer
Keywords: Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine; Paclitaxel

STUDY DESIGN:
Intervention Model Description: participants are randomized in a 2-1 fashion to Arm A vs. Arm B
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A. T-DM1 followed by Trastuzumab SC (Experimental): Randomized participants will receive intravenous T-DM1 every 3 weeks for 6 cycles (18 weeks) and then Trastuzumab SC (subcutaneous) every 3 weeks for 11 cycles
  Interventions: Drug: trastuzumab-emtansine; Drug: Trastuzumab SC
- Arm B: Paclitaxel with Trastuzumab SC, followed by Trastuzumab SC alone (Experimental): Randomized participants will receive weekly intravenous Paclitaxel for 12 weeks (4 cycles) and Trastuzumab SC (subcutaneous) every 3 weeks for 17 cycles. The first 4 doses Trastuzumab SC are given with Paclitaxel.
  Interventions: Drug: Trastuzumab SC; Drug: Paclitaxel

INTERVENTIONS:
Drug: trastuzumab-emtansine — intravenous infusion
  Other Names: T-DM1; Kadcyla
  Arms: Arm A. T-DM1 followed by Trastuzumab SC
Drug: Trastuzumab SC — Muscular injection
  Other Names: Herceptin Hylecta
Drug: Paclitaxel — intravenous infusion
  Other Names: Taxol; Onxal
  Arms: Arm B: Paclitaxel with Trastuzumab SC, followed by Trastuzumab SC alone

SUMMARY:
This research study is studying how well newly diagnosed breast cancer that has tested positive for a protein called HER2 responds using one of two different combination of HER2-directed therapies as a treatment after surgery.

The name of the study drugs involved are:

* Trastuzumab-emtansine (T-DM1, Kadcyla)
* Trastuzumab SC (Herceptin Hylecta)
* Paclitaxel

DETAILED DESCRIPTION:
This is a randomized phase II adjuvant study for women and men with Stage I HER2-positive invasive breast cancer. Participants will be randomized into one of two treatment arms in this study and receive:

* Arm 1: trastuzumab-emtansine (T-DM1, Kadcyla) and trastuzumab SC (Herceptin Hylecta)
* Arm 2: paclitaxel and trastuzumab SC (Herceptin Hylecta) This research study is looking to see if the study drug T-DM1 followed by trastuzumab SC will have less side-effects than traditional HER2-positive breast cancer treatment of trastuzumab and paclitaxel.The study is also looking to learn about the long-term benefits and disease-free survival of participants who are treated with T-DM1 followed by trastuzumab SC.

T-DM1 is an antibody-drug conjugate; it is made up of an antibody (trastuzumab) linked to a cytotoxic drug, DM1 (chemotherapy). T-DM1 functions as a targeted cancer therapy because it targets HER2-positive breast cancer cells directly, limiting exposure of the rest of the body to chemotherapy. More specifically, the trastuzumab in T-DM1 first binds to the HER2 protein on the surface of the breast cancer cells and the DM1 then enters the cells and can cause them to die, preventing tumor growth. The FDA (the U.S. Food and Drug Administration) has not approved T-DM1 for use on its own in patients with stage I, II, or III breast cancer. However, it has been approved for use in (a) advanced or metastatic, previously treated breast cancer and (b) in some patients receiving postoperative treatment after preoperative chemotherapy and surgery have been completed.

Trastuzumab SC is a subcutaneous form of trastuzumab.Trastuzumab is a monoclonal antibody, which are disease-fighting proteins made by cloned immune cells. Paclitaxel and trastuzumab are considered a standard-of-care regimen in early breast cancer. Trastuzumab is FDA-approved to be administered as an IV (intravenous) or subcutaneous (muscular injection).

The research study procedures include screening for eligibility and study treatment including laboratory evaluations and follow up visits.

Participants will receive study treatment for a year in total and will be followed for 5 years after treatment.

It is expected that about 500 people will take part in this research study.

Genentech is supporting this research study by providing funding for the study and supplying trastuzumab-emtansine (T-DM1) and trastuzumab SC (subcutaneous).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have HER2-positive Stage I histologically confirmed invasive carcinoma of the breast. Patients must have node-negative (N0) or micrometastases (N1mic) breast cancer according to the AJCC 8th edition anatomic staging table.

  * If the patient has had a negative sentinel node biopsy, then no further axillary dissection is required, and the patient is determined to be node-negative. If an axillary dissection without sentinel lymph node biopsy is performed to determine nodal status, at least six axillary lymph nodes must be removed and analyzed, and determined to be negative, for the patient to be considered node-negative. Axillary nodes with single cells or tumor clusters ≤ 0.2 mm by either H&E or immunohistochemistry (IHC) will be considered node-negative.
  * Any axillary lymph node with tumor clusters between 0.02 and 0.2 cm is considered a micrometastasis. Patients with a micrometastasis are eligible. An axillary dissection is not required to be performed in patients with a micrometastasis found by sentinel node evaluation. In cases where the specific pathologic size of lymph node involvement is subject to interpretation, the principal investigator will make the final determination as to eligibility. The investigator must document approval in the patient medical record.
  * Patients who have an area of a T1aN0, ER+ (defined as >10%), HER2-negative cancer in addition to their primary HER2-positive tumor are eligible.
* HER2-positive by ASCO CAP 2018 guidelines, confirmed by central testing. NOTE: HER-2 status must be confirmed to be positive by central review by NeoGenomics prior to patient starting protocol therapy. Patients previously having had HER2 immunohistochemical testing by NeoGenomics do not need to undergo retesting for central confirmation of HER2 status.

NOTE: DCIS components will not be counted in the determination of HER2 status

* ER/PR determination is required. ER and PR assays should be performed by immunohistochemical methods according to the local institution standard protocol.
* Bilateral breast cancers that individually meet eligibility criteria are allowed.
* Patients with multifocal or multicentric disease are eligible, as long as each tumor individually meets eligibility criteria. Central confirmation is needed for any site of disease that is tested to be HER2-positive by local testing (unless testing was previously done by NeoGenomics).
* Patients with a history of ipsilateral DCIS are eligible if they were treated with wide excision alone, without radiation therapy, or treated with a mastectomy for this current breast cancer. Patients with a history of contralateral DCIS are not eligible.
* ≤ 90 days between the planned treatment start date and the patient's most recent breast surgery for this breast cancer
* ≥ 18 years of age with any menopausal status.
* ECOG Performance Status 0 or 1
* All tumor should be removed by either a modified radical mastectomy or a segmental mastectomy (lumpectomy), with either a sentinel node biopsy or axillary dissection

  * All margins should be clear of invasive cancer or DCIS (i.e. no tumor on ink). The local pathologist must document negative margins of resection in the pathology report. If all other margins are clear, a positive posterior (deep) margin is permitted, provided the surgeon documents that the excision was performed down to the pectoral fascia and all tumor has been removed. Likewise, if all other margins are clear, a positive anterior (superficial; abutting skin) margin is permitted provided the surgeon documents that all tumor has been removed.
* Patients undergoing breast conservation therapy (i.e. lumpectomy) must not have any contraindications to radiation therapy. Radiation to the conserved breast is required.
* Patients may have received up to 4 weeks of tamoxifen therapy, or other hormonal therapy, for adjuvant therapy for this cancer. Patients cannot receive adjuvant hormonal therapy during protocol treatment for the first 12 weeks.
* Prior oophorectomy for cancer prevention is allowed.
* Patients who have undergone partial breast radiation (duration ≤ 14 days) prior to registration are eligible. Partial breast radiation must be completed prior to 2 weeks before starting protocol therapy. Patients who have undergone whole breast radiation are not eligible.
* Patients who have participated in a window study (treatment with an investigational agent prior to surgery for ≤ 2 weeks) are eligible. Patients must have discontinued the investigational agent at least 14 days before participation.
* Adequate bone marrow function:

  * ANC ≥ 1000/mm3,
  * Hemoglobin ≥ 9 g/dl
  * Platelets ≥ 100,000/mm3
* Adequate hepatic function:

  * Total bilirubin ≤ 1.2mg/dL
  * AST and ALT ≤ 1.5x Institutional ULN
  * For patients with Gilbert syndrome, the direct bilirubin should be within the institutional normal range. Serum alkaline phosphatase should be ≤ 1.5x Institutional ULN.
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Premenopausal patients must have a negative serum or urine pregnancy test, including women who have had a tubal ligation and for women less than 12 months after the onset of menopause.
* Women of childbearing potential and men with partners of childbearing potential must be willing to use one highly effective form of nonhormonal contraception or two effective forms of nonhormonal contraception by the patient and/or partner. Contraceptive use must be continued for the duration of the study treatment and for 7 months after the last dose of study treatment. Hormonal birth control methods are not permitted.
* Patients should have tumor tissue available, and a tissue block of sufficient size to make 15 slides, which must be sent to DFCI for correlative research. If a tissue block is unavailable, sites may send one H&E-stained slide and 15 unstained sections of paraffin-embedded tissue on uncharged slides. Slide sections should be 4-5 microns in thickness. It is also acceptable to submit 2 cores from a block of invasive tissue using a 1.2 mm diameter coring tool. If tumor is not available, the investigator must document why tissue is not available in the patient medical record, and that efforts have been made to obtain tissue.
* Willing and able to sign informed consent
* Must be able to read and understand English in order to participate in the quality of life surveys. If patient does not read and understand English, the patient is still eligible, but cannot participate in the quality of life surveys.

Exclusion Criteria:

* Any of the following due to teratogenic potential of the study drugs:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragms, IUDs, surgical sterilization, abstinence, etc.).
  * Men who are unwilling to employ adequate contraception (condoms, surgical sterilization, abstinence, etc.).
* Locally advanced tumors at diagnosis, including tumors fixed to the chest wall, peau d'orange, skin ulcerations/nodules, or clinical inflammatory changes (diffuse brawny cutaneous induration with an erysipeloid edge)
* Patients with a history of previous invasive breast cancer.
* History of prior chemotherapy in the past 5 years.
* History of paclitaxel therapy
* Patients with active liver disease, for example due to hepatitis B virus, hepatitis C virus, autoimmune hepatic disorder, or sclerosing cholangitis
* Individuals with a history of a different malignancy are ineligible except for the following circumstances:

  * Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy.
  * Individuals with the following cancer are eligible regardless of when they were diagnosed and treated: cervical cancer in situ, and non-melanoma cancer of the skin.
* Intercurrent illness including, but not limited to: ongoing or active, unresolved systemic infection, renal failure requiring dialysis, active cardiac disease, prior myocardial infarction (asymptomatic changes on EKG suggestive of old MI is not an exclusion), history of CHF, current use of any therapy specifically for CHF, uncontrolled hypertension, significant psychiatric illness, or other conditions that in the opinion of the investigator limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinically relevant toxicities (CRT) | First 18 weeks of treatment
  Compare the incidence of clinically relevant toxicities (CRT) in patients with Stage I HER2-positive breast cancer treated with trastuzumab emtansine followed by trastuzumab SC to the incidence in those treated with paclitaxel in combination with trastuzumab SC as assessed by PRO-CTCAE
Disease Free Survival (DFS) | Time from randomization to first Disease Free Survival (DFS) event up to 72 months
  Evaluate disease-free survival in the T-DM1 followed by trastuzumab SC arm

SECONDARY OUTCOMES:
Grade 3 and 4 adverse events | Enrollment to end of treatment up to 1 year
  Compare the incidence of all grade 3 and 4 adverse events in patients treated with adjuvant trastuzumab emtansine followed by trastuzumab SC to the incidence in those receiving paclitaxel in combination with trastuzumab SC
Quality of Life Assessment: FACT B | Enrollment to end of treatment up to 1 year
  Compare responses to FACT-B quality of life (QOL) questionnaire in patients receiving trastuzumab emtansine followed by trastuzumab SC to that experienced by patients receiving paclitaxel in combination with trastuzumab SC.
Symptoms related to therapy | Enrollment to end of treatment up to 1 year
  Evaluate symptoms related to therapy in patients receiving trastuzumab emtansine followed by trastuzumab SC compared to those receiving paclitaxel in combination with trastuzumab SC using the Rotterdam Symptom Checklist (RSCL)
Symptoms related to therapy | Enrollment to end of treatment up to 1 year
  Evaluate symptoms related to therapy in patients receiving trastuzumab emtansine followed by trastuzumab SC compared to those receiving paclitaxel in combination with trastuzumab SC using the Patient Neurotoxicity Questionnaire (PNQ)
Effects of therapy on work productivity | Enrollment to end of treatment up to 1 year
  Evaluate effects of therapy on work productivity and activity using the Work Productivity and Activity Impairment Questionnaire (WPAI-SHP) in patients receiving trastuzumab emtansine followed by trastuzumab SC compared to those receiving paclitaxel in combination with trastuzumab SC
Effect of alopecia on patients | Enrollment to end of treatment up to 1 year
  Evaluate the effects of alopecia on patients receiving paclitaxel in combination with trastuzumab SC using an alopecia questionnaire
Incidence of Side Effects | Enrollment to end of treatment up to 1 year
  Compare incidence of sensory neuropathy, headache, arthralgia and myalgia using PRO-CTCAE criteria in patients receiving trastuzumab emtansine followed by trastuzumab SC to that experienced by patients receiving paclitaxel in combination with trastuzumab SC
Incidence of grade 3-4 cardiac left ventricular dysfunction | Enrollment to end of treatment up to 1 year
  Evaluate the incidence of grade 3-4 cardiac left ventricular dysfunction in patients treated with adjuvant trastuzumab emtansine followed by trastuzumab SC compared to those receiving paclitaxel with trastuzumab SC
Incidence of trastuzumab-emtansine-induced grade 2-4 thrombocytopenia | Enrollment to end of treatment up to 1 year
  Evaluate the incidence of trastuzumab-emtansine-induced grade 2-4 thrombocytopenia
Percentage of patients with amenorrhea | Enrollment to end of treatment up to 1 year
  Investigate the percentage of patients with amenorrhea at various time points after the start of treatment in premenopausal women receiving treatment with trastuzumab emtansine followed by trastuzumab SC and paclitaxel with trastuzumab SC
Evaluation of gene predictors of trastuzumab-emtansine-induced grade 2-4 | Enrollment to end of treatment up to 1 year
  Evaluate gene biomarkers predictive of trastuzumab-emtansine-induced grade 2-4 thrombocytopenia
Gene Profiling | Enrollment to end of treatment up to 1 year
  Utilize genomic profiling to query a large panel of cancer gene mutations and gene expression in patients with Stage I HER2-positive breast cancer
Radiation therapy Toxicity | Enrollment to end of treatment up to 1 year
  Evaluate the incidence of toxicities attributed to radiation therapy when given concurrently with trastuzumab SC after receipt of either trastuzumab emtansine or paclitaxel
Overall survival | Enrollment to end of treatment up to 1 year
  Describe overall survival in patients with Stage I HER2-positive breast cancer treated with trastuzumab emtansine followed by trastuzumab SC

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (51):
- United States (51):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Smilow Cancer Hospital Care center at Derby, Derby, Connecticut
  - Smilow Cancer Hospital Care center at Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care center at Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care center at St. Francis, Hartford, Connecticut
  - Smilow Cancer Hospital Care center at Long Ridge, Long Ridge, Connecticut
  - Yale Cancer Center at Yale University School of Medicine, New Haven, Connecticut
  - Smilow Cancer Hospital Care center at North Haven, North Haven, Connecticut
  - Stamford Hospital, Stamford, Connecticut
  - Smilow Cancer Hospital Care center at Torrington, Torrington, Connecticut
  - Smilow Cancer Hospital Care center at Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care center at Waterbury, Waterbury, Connecticut
  - Smilow Cancer Hospital Care center at Waterford, Waterford, Connecticut
  - Miami Cancer Institute/Baptist Hospital of Miami, Miami, Florida
  - Miami Cancer Institute - Plantation (MCIP), Plantation, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Health Joe & Shelly Schwarz Cancer Center, Carmel, Indiana
  - IU Health North Hospital, Carmel, Indiana
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Indiana University Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Eastern Maine Medical Center (Northern Light), Brewer, Maine
  - New England Cancer Specialists, Scarborough, Maine
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber at St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Mass General North Shore Cancer Center, Danvers, Massachusetts
  - Dana-Farber Brigham Cancer Center - Foxborough, Foxborough, Massachusetts
  - Dana-Farber Cancer Instiute - Merrimack Valley, Methuen, Massachusetts
  - Dana-Farber at Milford, Milford, Massachusetts
  - Newton Wellesley Hospital, Newton, Massachusetts
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Dana Farber at South Shore Hospital, Weymouth, Massachusetts
  - NH Oncology-Hematology, PA - Payson Center for Cancer Care, Concord, New Hampshire
  - Dana-Farber Cancer Insitute at Londonderry Hospital, Londonderry, New Hampshire
  - Solinsky Center for Cancer Care (NH Oncology-Hematology, PA), Manchester, New Hampshire
  - New England Cancer Specialists - Portsmouth, Portsmouth, New Hampshire
  - New York University Langone Hospital -Brooklyn, Brooklyn, New York
  - New York University Langone Hospital - Long Island, Mineola, New York
  - New York University Langone Health, New York, New York
  - Northwell University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Stefanie Spielman Comprehensive Breast Center, Columbus, Ohio
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Smilow Cancer Hospital Care center at Westerly, Westerly, Rhode Island
  - Greco-Hainsworth Centers for Research/Tennessee Oncology, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu